CLINICAL TRIAL: NCT03504553
Title: The Effect of a Reduced Noise Environment on Induction and Emergence Behavior in Children Undergoing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joshua Uffman (Other)
Responsible Party: Sponsor-Investigator, Joshua Uffman, Vice Chair, Department of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-00203
Record Dates: First submitted 2018-04-12; First posted 2018-04-20 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Surgery; Noise Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noise reduction (Experimental): Reduced operating room personnel, low ambient light and soft background music during induction and emergence from anesthesia.
  Interventions: Other: Noise reduction
- Control (No Intervention): Normal operating room environment.

INTERVENTIONS:
Other: Noise reduction — All activity will cease when the patient enters the operating room and nonessential personnel will be removed. Ambient lighting will be reduced and communication devices muted.
  Arms: Noise reduction

SUMMARY:
This project will investigate whether reduction in ambient light and elimination of noise on induction of anesthesia alters anxiety (modified Yale Preoperative Anxiety Scale or mYPAS) or compliance (induction compliance checklist or ICC scoring), alters recovery following emergence using pain scores, analgesic requirements, and emergence delirium (post anesthesia emergence delirium or PAED), or post-discharge behavior at 1, 7 and 14 days (modified post hospitalization behaviour questionnaire or PHBQ) in patients who receive anxiolytic premedication. In addition, the investigators will assess the cumulative level of nose exposure that patients experience during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing general anesthesia for tonsillectomy/adenoidectomy, tympanomastoidectomy, or general abdominal laparoscopic surgical procedures lasting at least 30 minutes.
* Receiving midazolam prior to the procedure as part of standard of care.

Exclusion Criteria:

* Patients that are taking antidepressant medications, anxiolytic medication, analgesia medications other than acetaminophen or NSAIDs.
* Allergy to midazolam.
* History of emergence delirium.
* Cardiac disease, other than functional heart murmurs.
* Developmental delays.
* Parent refusal of midazolam for standard clinical care.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2018-10-18 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Anxiety during induction | First 5 minutes of surgical procedure
  A blinded observer will assess behavior prior to and during induction/placement of face mask or insertion of an intravenous line using the mYPAS scale.

SECONDARY OUTCOMES:
Compliance during induction | First 5 minutes of surgical procedure
  A blinded observer will assess behavior prior to and during induction/placement of face mask or insertion of an intravenous line using the ICC scale.
Presence of post anesthesia emergence delirium | Average of 30 mins - 1 hr
  Following transfer to the post anesthesia care unit (PACU) from the OR, the PAED scale will be measured every 10 minutes from arrival until discharge from PACU.
Post-discharge behavior disturbances | Post-op day 1
  Parents will be contacted by phone and asked a series of 11 questions (PHBQ) to assess participants behavior following surgery.
Post-discharge behavior disturbances | Post-op day 2
  Parents will be contacted by phone and asked a series of 11 questions (PHBQ) to assess participants behavior following surgery.
Post-discharge behavior disturbances | Post-op day 7
  Parents will be contacted by phone and asked a series of 11 questions (PHBQ) to assess participants behavior following surgery.
Noise exposure | Average of 30 mins - 3 hrs
  Assess the peak and cumulative level of noise exposure to the patient during the entire surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cartabuke, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Bozych M, Tram NK, Rice-Weimer J, Cartabuke RS, Tobias JD, Huffman J, Mpody C, Uffman JC. Operating Room Noise Environment and Behavior in Children Undergoing General Anesthesia: A Randomized Controlled Trial. Anesthesiol Res Pract. 2024 Aug 16;2024:4838649. doi: 10.1155/2024/4838649. eCollection 2024. PMID 39185368